CLINICAL TRIAL: NCT07389018
Title: Prospective Longitudinal Monocentric Study to Evaluate the Feasibility of Syde® Digital Endpoints for Monitoring Patients With Progressive Supranuclear Palsy - Richardson Syndrome (PSP-R)
Acronym: PROSPER-SYDE
Status: Not yet recruiting | Type: Observational
Sponsor: SYSNAV (Industry)
Responsible Party: Sponsor
Other Study IDs: PR5030-76; 2024-A02611-46 (Other: ANSM)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Progressive Supranuclear Palsy- Richardson Syndrome (PSP-R)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess the feasibility/acceptability of real-world activity monitoring by the Syde® wearable device in PSP-R. The Syde® collected data will be compared to on-site conventional clinical endpoints, including functional capacity and cognitive assessments, as well as core scales assessments.

ELIGIBILITY:
Inclusion Criteria:

1.18 years old or older

2.Participants affiliated to, or beneficiary from, a social security.

3.Ambulant patients (i.e. able to walk 10 meters without assistance)

4.Signed informed consent form by the patient himself or, by caregivers if the patient is not capable to fill, date and sign the form due to fine motor function difficulties..

5.Possible or probable PSP-R according to MDS criteria 2017(Hoglinger et al., Mov Disorder, 2017).

Exclusion Criteria:

1. Patients with extreme cognitive disorders that limit their understanding of the data collection process (training of device use and 4-week recording periods every 4 months, device return at the end of the study), tests to be performed including eye movement recording (every 8 months), the implication of the study and consent.
2. Patients who do not tolerate to keep the sensors on their ankles.
3. Patients who have undergone a surgical procedure or who have experienced recent trauma (within fewer than 6 months) affecting the lower limbs.
4. A concomitant chronic or acute neurological, endocrine, infectious, allergic, or inflammatory pathology within the 3-week period immediately prior to inclusion.
5. Patients affected by any other disorder having a significant impact on gait or lower limb function.
6. Participant covered by a legal protection measure (guardianship, curatorship or safeguarding of justice) or who is unable to express their consent.
7. Absence of caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Progressive Supranuclear Palsy - Richardson Syndrome (PSP-R)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients reaching the optimal threshold of recordings during the recording periods defined in the protocol. | 16 months
  Number of patients reaching the optimal threshold of recordings during the recording periods defined in the protocol (supposed optimal threshold for analysis) at baseline, Month 4, Month 8, Month 12 and Month 16.
Usability score at Month 4 and at the end of the study | 16 months
  Usability score at Month 4 and Month 16

SECONDARY OUTCOMES:
Change from baseline in the total wearing time at months 4, 8, 12, and 16. | 16 months
  Change from baseline in the total wearing time at months 4, 8, 12, and 16.
Reproducibility for each recording period timepoint | 16 months
  Reproducibility assessed by the ICC (Intra-Class Correlation) and Bland and Altman analysis for each recording period timepoint (baseline, 4 months, 8 months, 12 months, and 16 months)
Correlation between Syde® digital endpoints and 2-minute walk test (2MWT) | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and 2MWT
Correlation between Syde® digital endpoints and 10-meter walk test (10MWT) | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and 10MWT
Correlation between Syde® digital endpoints and Timed Up and Go (TUG) | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and TUG
Correlation between Syde® digital endpoints and falls reported by the participants | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and falls reported by the participants
Correlation between Syde® digital endpoints and Progressive Supranuclear Palsy Rating Scale (PSP-RS) | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and PSP-RS
Correlation between Syde® digital endpoints and Progressive Supranuclear Palsy Clinical Deficits Scale (PSP-CDS) | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and PSP-CDS
Correlation between Syde® digital endpoints and Montreal Cognitive Assessment (MoCA) | 16 months
  Correlation at baseline and at different timepoints between Syde® digital endpoints and MoCA
Longitudinal change in Syde® digital endpoints. The Syde® digital endpoints will include the SV95C (Stride Velocity 95th centile) | 16 months
  Change from baseline in Syde® digital endpoints at 4, 8, 12 and 16 months. The Syde® digital endpoints will include the SV95C (Stride Velocity 95th centile)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe BRANDEL, Principal Investigator — Hopital Fondation Adolphe de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France